CLINICAL TRIAL: NCT05425108
Title: Effectiveness of Binocular Peripheral Myopic Projected Defocus on Ocular Biometrics Using a Clinical Prototype Device
Brief Title: Binocular Peripheral Myopic Defocus Using a Clinical Prototype Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kubota Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP1 Pilot
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- CP1 device (Active Comparator)
  Interventions: Device: Binocular CP1
- Control (No Intervention)

INTERVENTIONS:
Device: Binocular CP1 — Binocular active projection of defocused image in the peripheral visual field
  Arms: CP1 device

SUMMARY:
Kubota Vision Inc. has developed a spectacle-like prototype device which is designed to be used as a light-based therapy to reduce myopia progression. In this study, we aim to observe the ocular biometric and refractive changes following binocular part-time wear of the clinical prototype device over a course of 12 months and compare that to 12 months of no clinical prototype device use (control).

ELIGIBILITY:
Inclusion Criteria:

* Spherical equivalent -0.50 to -5.50 diopters
* visual acuity of at least 20/25 in each eye

Exclusion Criteria:

* history of ocular trauma or major eye surgery
* active ocular infection
* any prior history or participation in myopia control treatments within the past 3 months

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Central axial length | 12 months
Cycloplegic refraction | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arkady Selenow, OD, Principal Investigator — Manhattan Vision Associates/Institute of Vision Research
Locations (1):
- Manhattan Vision Associates/Institute of Vision Research, New York, New York, United States